CLINICAL TRIAL: NCT06066970
Title: Cardiac Biomarkers for the Quantification of Myocardial Damage After Cardiac Surgery
Acronym: RORSCHACH
Status: Recruiting | Type: Observational
Sponsor: Jena University Hospital (Other)
Responsible Party: Principal Investigator, Tulio Caldonazo, Principal Investigator, Jena University Hospital
Other Study IDs: ZKSJ0156
Record Dates: First submitted 2023-09-28; First posted 2023-10-04 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Cardiac Valve Disease
Keywords: Biomarker; Troponin; CK-MB; Perioperative Myocardial Infarction; LGE-cMRI
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sampling - analysis of cardiac biomarker release (Troponin I, Troponin T, CK-MB, CK).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of the study is to clarify whether the perioperative release of the cardiac biomarkers troponin I, troponin T and CK-MB consistently correlate with visualizable myocardial damage, and to what extent these biomarkers are comparable by means of their kinetics and dynamics.

Due to the uncertainty regarding the validity of cardiac biomarkers in the diagnosis of myocardial infarction, the answer to these questions could have a considerable influence on internationally valid guidelines and definitions. International studies, especially in the field of coronary surgery and coronary artery disease treatment refer to these definitions, in particular, the adequate treatment of affected patients is directly dependent on them.

DETAILED DESCRIPTION:
In the course of a myocardial infarction, the death of cardiomyocytes leads to the release of specific cardiac biomarkers (CK-MB, troponin I and T). Since there is a general risk of perioperative infarction in cardiac surgery, the standard monitoring includes appropriate diagnostics. These are based on clinical symptoms, ECG, imaging (echocardiography or coronary angiography) and, in particular, the elevation of these cardiac biomarkers. Recently, the latter have been regularly moved into the foreground as the sole indicators of perioperative myocardial infarction, and first definitions allow the diagnosis solely based on troponin or CK-MB elevation.

However, biomarker elevations may not be accompanied by an image-morphologically detectable perfusion defect (myocardial infarction). Such phenomena have been described outside of cardiac surgery, for example, in marathon runners4, but also due to comorbidities such as renal insufficiency or neurological diseases. Even in patients undergoing cardiac surgery without coronary artery disease (e.g., isolated valve surgery), biomarker elevations up to the infarct-defining range are regularly observed. Whether in the latter case the perioperative routinely observed troponin or CK-MB elevation are indeed related to surgery-induced chronic perfusion disturbance has not yet been investigated.

To date, there is no study that quantitatively correlates purely perioperatively induced ischemic damage with the release of cardiac biomarkers. In addition, the three most commonly used biomarkers for perioperative infarct diagnosis differ considerably in their temporal release and release dynamics. Moreover, a direct comparison of all three parameters has never been performed so far.

Therefore, the aim of this study is to quantify and compare the release of troponin T, I and CK/CK-MB in the postoperative course in patients without relevant coronary artery disease undergoing elective isolated heart valve surgery. These findings will subsequently be correlated with classical diagnostics (clinic, ECG, echocardiography) and image morphological quantification of perioperatively induced myocardial damage by magnetic resonance imaging (LGE-cMRI).

ELIGIBILITY:
Inclusion Criteria:

* Indication for isolated aortic or mitral valve surgery
* Written informed consent
* Age ≥ 18 years

Exclusion Criteria:

* Presence of coronary artery disease (excluded within the last 6 months)
* Allergy to gadolinium
* Cochlear implant
* Deep brain stimulation
* Individual factors excluding the performance of an MRI (e.g. claustrophobia of the patient)
* Significantly reduced renal function (GFR < 30ml/min)
* Perioperative complications that may lead to myocardial damage (discontinuation of the study for the patient and exclusion from the analysis after primary study inclusion)
* Need for extension of surgery (additional procedures on other heart valves, aorta, myocardium, or similar; exclusion after primary study inclusion possible)
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indication for isolated aortic or mitral valve surgery and exclusion of coronary artery disease.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation biomarker release and LGE-cMRI | pre-surgery and 5 days post-surgery
  Correlation of the peak value of the respective biomarker with the amount of perioperatively induced myocardial damage quantified by LGE-cMRI.

CONTACTS AND LOCATIONS:
Overall Officials: Tulio Caldonazo, Dr., Principal Investigator — Jena University Hospital
Locations (5):
- Germany (5):
  - Universitäts-Herzzentrum Freiburg • Bad Krozingen, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitätsklinikum Halle, Halle, Saxony-Anhalt
  - Universitätsklinikum Jena, Jena, Thuringia

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet decided in which way and which data exactly will be shared with other researchers.

REFERENCES:
- [Derived] Caldonazo T, Winter M, Kiehntopf M, Aschenbach R, Grager S, Reinartz S, Scherag A, Schumacher U, Kirov H, Teichgraber U, Doenst T; RORSCHACH Investigators and GermaN HeaRTS. Cardiac biomarkers for the quantification of myocardial damage after cardiac surgery - The RORSCHACH trial. Int J Cardiol Heart Vasc. 2025 Aug 28;60:101781. doi: 10.1016/j.ijcha.2025.101781. eCollection 2025 Oct. PMID 40918750